CLINICAL TRIAL: NCT06502977
Title: Phase 2a Study Evaluating the Efficacy, Safety, Tolerability and Pharmacokinetics of Tarlatamab in Chinese Subjects With Advanced Small Cell Lung Cancer After Two or More Prior Lines of Treatment (DeLLphi-307)
Brief Title: Study Evaluating Tarlatamab in Chinese Participants With Advanced Small Cell Lung Cancer After Two or More Prior Lines of Treatment
Acronym: DeLLphi-307
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230273
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Extensive Stage Small Cell Lung Cancer; Advanced Small Cell Lung Cancer; SCLC; AMG 757; Tarlatamab; IMDELLTRA; Tumor; Programmed Cell Death Protein 1; Programmed Cell Death Ligand 1; PD-1 Protein; PD-L1 Protein; Pharmacokinetics; Malignancy; Cancer; Chinese Participants; China; Platinum; Platinum-based; Neuroendocrine tumor; Bi-specific T-cell engager; BiTE molecule
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors | interventions — AMG 757

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tarlatamab (Experimental): Participants will receive tarlatamab as an intravenous (IV) infusions in 28-day cycles.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — IV infusion
  Other Names: AMG 757; IMDELLTRA™

SUMMARY:
The primary aim of this study is to evaluate the efficacy of tarlatamab as assessed by objective response rate (ORR) based on blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Participant must be a resident in China, and of Chinese ancestry ≥ 18 years of age (or legal adult age within country) at the time of signing the informed consent.
* Histologically or cytologically confirmed small cell lung cancer.
* Extensive-stage SCLC participants who progressed on or recurred following 1 platinum-based regimen as 1L therapy (including a PD-1/PD-[L]1) and at least 1 other prior line of therapy.
* Measurable lesions as defined per RECIST 1.1 within 21 days prior to the first dose of study drug.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Minimum life expectancy of 12 weeks.
* Adequate organ function.

Exclusion Criteria:

Disease Related

* Any previous diagnosis of transformed non-small cell lung cancer (NSCLC), epidermal growth factor receptor (EGFR) activating mutation positive NSCLC that has transformed to SCLC.
* Symptomatic central nervous system (CNS) metastases.
* Diagnosis or evidence of leptomeningeal disease.
* Prior history of severe or life-threatening events from any immune-mediated therapy.

Other Medical Conditions

* Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
* History of solid organ transplantation.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of other malignancy within the past 2 years, with certain exceptions
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of study drug.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of first dose of study drug.
* Participants with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study drug.
* HIV, Hepatitis B, and Hepatitis C, with certain exceptions.
* Major surgery within 28 days of first dose study drug. Prior/Concomitant Therapy
* Currently or previously enrolled in a tarlatamab study.
* Prior therapy with any selective inhibitor of the DLL3 pathway.
* Prior anti-cancer therapy within 21 days prior to first dose of study treatment, with certain exceptions.
* Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug, with certain exceptions.
* Treatment with live virus, including live-attenuated vaccination, within 14 days prior to the first dose of study drug. Inactive vaccines (eg, non-live or non-replicating agent) and live viral non-replicating vaccines (eg, Jynneos for mpox infection) within 3 days prior to first dose of study drug.

Prior/Concurrent Clinical Study Experience

• Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions

* Female participants of childbearing potential unwilling to use protocol-specified method of contraception during treatment and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Female participants who are breastfeeding or who plan to breastfeed while on study and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Female participants planning to become pregnant or donate eggs while on study and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional period of time after the last dose of study drug as specified in the study protocol.
* Participants has known sensitivity to any of the products or components to be administered during dosing.
* Participants likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures.
* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or medical monitor if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
ORR Based on BICR per RECIST 1.1 | Approximately 24 months

SECONDARY OUTCOMES:
Duration of Response (DOR) Based on BICR per RECIST 1.1 | Approximately 24 months
Disease Control (DC) Based on BICR per RECIST 1.1 | Approximately 24 months
Duration of DC Based on BICR per RECIST 1.1 | Approximately 24 months
Progression-free Survival (PFS) Based on BICR per RECIST 1.1 | Approximately 24 months
ORR Based on Investigator Assessment per RECIST 1.1 | Approximately 24 months
DOR Based on Investigator Assessment per RECIST 1.1 | Approximately 24 months
DC Based on Investigator Assessment per RECIST 1.1 | Approximately 24 months
Duration of DC Based on Investigator Assessment per RECIST 1.1 | Approximately 24 months
PFS Based on Investigator Assessment per RECIST 1.1 | Approximately 24 months
Overall Survival (OS) | Approximately 24 months
Number of Participants Who Experience Treatment-emergent Adverse Events (TEAEs) | Approximately 24 months
Serum Concentration of Tarlatamab | Approximately 24 months
Number of Participants with Anti-tarlatamab Antibody Formation | Approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Army Medical University, People's Liberation Army, Chongqing, Chongqing Municipality
  - Army Special Medical Center of Peoples Liberation Army, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Harbin Meidical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Fujian Cancer Hospital, Fuzhou

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com